CLINICAL TRIAL: NCT06911346
Title: Exploring the Role of Native Plant-Based Foods and (Poly)Phenol Supplementation in Modifying Gut-Microbiota Metabolism: A Strategy for Reducing Body Weight and Cardiometabolic Risk
Brief Title: Plant-Based Foods and (Poly)Phenol Supplementation in Gut Microbiota Modulation, Body Weight, and Cardiometabolic Risk
Acronym: PREDIET-ARAC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Catolica de Temuco (Other)
Collaborators: Agencia Nacional de Investigación y Desarrollo (Other)
Responsible Party: Principal Investigator, Dr. Fabián Ignacio Lanuza Rilling, Principal Investigator, Universidad Catolica de Temuco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Universidad Catolica de Temuco; FONDECYT Iniciación 11250095 (Other Grant/Funding Number: Chilean National Agency for Research and Development (ANID))
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-08

CONDITIONS: Obesity and Overweight
Keywords: Plant-Based Diet; Polyphenol Supplementation; Cardiometabolic Risk; Weight Loss; Gut Microbiota
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Who Masked: Participant
Masking Description: In addition to participant masking, investigators and outcome assessors will remain blinded to group assignments. Only the principal investigator will have access to the allocation information, while the rest of the research team will identify participants by ID only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dietary Supplementation Group (Experimental): Healthy plant-based diet (plus supplemental foods) as part of a hypocaloric diet.
  Interventions: Dietary Supplement: Diet supplementation
- Polyphenol-rich Supplement Group (Experimental): Hypocaloric diet with polyphenol-rich supplement.
  Interventions: Dietary Supplement: Polyphenol-rich supplement
- Placebo Control Group (Placebo Comparator): Hypocaloric diet plus Placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Diet supplementation — Healthy plant-based diet (plus supplemental foods) as part of a hypocaloric diet.
  Arms: Dietary Supplementation Group
Dietary Supplement: Polyphenol-rich supplement — Hypocaloric diet with polyphenol-rich supplement. Polyphenol-rich sachets containing ≈30g/day of a combination of plant extracts rich in polyphenol. Frequency: 2 sachets a day. Duration: 12 weeks
  Arms: Polyphenol-rich Supplement Group
Other: Placebo — Hypocaloric diet plus Placebo. The placebo is a sachet (≈30g/day) with similar appearance, taste, and texture but without active polyphenols. Frequency: 2 sachets a day. Duration: 12 weeks
  Arms: Placebo Control Group

SUMMARY:
This single-blind, randomized controlled trial aims to evaluate the effects of increased dietary polyphenol intake-either through a healthy plant-based diet (PBD) or supplementation-on body weight and cardiometabolic risk factors in adults with overweight or obesity.

A total of 99 participants (aged 25-45 years, BMI 25-35 kg/m²) with cardiovascular risk factors will be recruited from local health centers and randomly assigned (1:1:1) to one of three intervention groups for 12 weeks: (1) a healthy PBD rich in polyphenols, with supplemental apple, blueberries, hazelnuts, extra-virgin olive oil, and coffee provided at no cost to the participant (2) a healthy diet plus polyphenol supplementation (≈30g/day) from maqui , green tea, olive leaf, cranberry, and grape extracts, or (3) a control group receiving placebo and standard healthy diet recommendations. All groups will follow a caloric deficit.

Dietary intake will be assessed using three 24-hour dietary recalls at baseline and 12 weeks, with polyphenol intake estimated via the Phenol-Explorer database. Data collection will include lifestyle questionnaires, anthropometric and bioimpedance measurements, blood pressure assessments, physical activity monitoring via accelerometers, and strength evaluations. Blood samples will be analyzed using a large-scale targeted metabolomics approach (UHPLC-MS/MS) to identify metabolic signatures, particularly those linked to gut microbiota. Faecal samples will be collected at baseline and visit 3.

Findings will provide insights into how dietary polyphenols-either from whole foods or supplementation-affect obesity-related outcomes and cardiometabolic risk, potentially unveiling gut microbial biomarkers as future therapeutic targets. This study aims to contribute to strategies for obesity and cardiometabolic risk prevention and treatment.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the impact of increased dietary polyphenol intake-either through a healthy plant-based diet (PBD) or supplementation-on body weight and cardiometabolic risk factors in adults with overweight or obesity. Additionally, the study seeks to explore the role of gut-microbiota-derived metabolites as potential mediators of these effects through metabolomic analyses.

The calculation determined a required sample size of 90 participants. To account for potential dropouts, a 10% buffer was added, resulting in a final target of 99 participants (33 per group); trial power of 0.8 and alfa error of 5%. A total of 99 participants (aged 25-45 years, BMI 25-35 kg/m²) with at least three cardiometabolic risk factors will be recruited from Health Centers supported by the Health Department of the Municipality in Temuco, Chile.

Participants will be randomly assigned (stratified by sex and age: <35y and ≥35y) in a 1:1:1 ratio to one of three groups for a 12-week intervention, with assessments conducted at baseline, week 6, and week 12:(1) a group following a healthy PBD rich in polyphenols, (2) a group following a healthy diet plus polyphenol supplementation (≈30g/day from maqui, green tea, cranberry, olive leaf and grape extracts), and (3) a control group receiving placebo and standard dietary recommendations. All groups will follow a caloric deficit (~1,200 kcal/day) for the entire 12-week study. This will be explained to each participant during the first visit.

Dietary data will be collected using three 24-hour dietary recalls at baseline and after 12 weeks, employing the SER 24 HDR software. The SER-24H software (University of Chile; Santiago, Chile) developed by CIAPEC (Center for Research in Food Environments and Prevention of Nutrition-Associated Diseases) at INTA, University of Chile, was used for dietary assessment. The Phenol-Explorer database estimates dietary polyphenol intake. It is the first comprehensive database on polyphenol content in foods. It contains more than 35,000 content values for 500 different polyphenols in over 400 foods.

Lifestyle, general health, and physical activity will be assessed through validated questionnaires. Anthropometric and body composition measurements will be taken using bioimpedance analysis. Blood pressure will be monitored with sphygmomanometers, while muscle strength will be measured via dynamometry.

Biological samples, including blood and plasma, will be collected at baseline and after 12 weeks. On each visit, 20ml of blood will be extracted from the antecubital vein and will be centrifuged and stored at -80ºC in the ultra-freezers of the School of Medicine at the Catholic University of Temuco until used.

Additionally, participants will be invited to provide a faecal sample during the first and third visits. These samples are not part of the main study but will be stored at -80ºC for potential future microbiota analyses (School of Medicine at the Catholic University of Temuco).

Biochemical analyses will be performed by institutional laboratory. Blood tests will include rutinary hematology and biochemistry, and inflammatory parameters.

Targeted metabolomic analyses will be conducted using ultra-high performance liquid chromatography coupled to tandem mass spectrometry (UHPLC-MS/MS) to identify and quantify polyphenol-derived metabolites, gut microbial metabolites, and other biochemical markers relevant to obesity and cardiometabolic risk.

Participants in the PBD group will receive a structured dietary plan featuring regional and national polyphenol-rich foods such as blueberries, hazelnuts, olive oil, apples, and coffee. The polyphenol supplementation group will receive a standardized supplement taken twice daily. The control group will receive placebo and standard nutritional counseling.

The study will adhere to ethical guidelines, including the Declaration of Helsinki and Good Clinical Practice principles. Ethical approval will be obtained, and all participants will provide informed consent. Data privacy will be ensured in compliance with applicable regulations.

Statistical analyses will be conducted on an intention-to-treat and per-protocol basis. Primary outcomes include changes in body weight and body composition, while secondary outcomes focus on cardiometabolic risk factors, dietary adherence, and metabolic signatures identified through metabolomics. Differences between pre- and post-intervention data, as well as between groups, will be analyzed using multivariate models, machine-learning algorithms, and generalized linear mixed models (GLMMs).

ELIGIBILITY:
Inclusion Criteria:

* Age between 25 and 45 years (adult)
* Sexes: All
* Overweight or obesity class I (BMI 25-35 kg/m²)
* At least three of the following cardiometabolic risk factors:

Current smoker (more than 1 cigarette per day during the last month) Sitting time greater than 7 hours per day or classified as inactive according to the IPAQ Fasting glucose ≥100 mg/dL (5.6 mmol/L)

High blood pressure:

Systolic blood pressure >130 mmHg Diastolic blood pressure >85 mmHg High serum triglycerides (≥150 mg/dL) HbA1c ≥38 mmol/mol (>5.7%)

Waist circumference defined by Peterman et al. for the Chilean population:

92.3 cm for men 87.6 cm for women High high-sensitivity C-reactive protein (hs-CRP) (≥2.0 mg/L)

Family history of premature coronary heart disease:

Definite myocardial infarction or sudden death before age 55 in father or male first-degree relative Before age 65 in mother or female first-degree relative

Exclusion Criteria:

* Presence of cardiovascular disease, diabetes, or hypertension
* Severe medical conditions that may impair participation in a nutrition intervention study (e.g., digestive disease, advanced malignancy, major neurological or psychiatric disease)
* Any medical condition limiting survival to less than one year
* Illegal drug use, chronic alcoholism, or problematic alcohol use
* BMI ≥35 kg/m²
* Antibiotic use within the last month
* Low predicted likelihood of changing dietary habits according to the Prochaska and DiClemente stages of change model

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-06-03 (Estimated); Study Completion 2026-06-03 (Estimated)

PRIMARY OUTCOMES:
Body weight | Visit 1 (Baseline), Visit 2 (Week 6), Visit 3 (Week 12)
  Unit: Kilograms Measured with: bioimpedance scan

SECONDARY OUTCOMES:
Systolic blood pressure | Visit 1 (Baseline), Visit 2 (Week 6), Visit 3 (Week 12)
  Unit: mmHg Measured with: Sphygmomanometer
Diastolic blood pressure | Visit 1 (Baseline), Visit 2 (Week 6), Visit 3 (Week 12)
  Unit: mmHg Measured with: Sphygmomanometer
Glucose | Visit 1 (Baseline), Visit 3 (Week 12)
  Plasma concentrations (mg/dl)
Glycosylated hemoglobin | Visit 1 (Baseline), Visit 3 (Week 12)
  Measured through plasma concentrations Unit: %
Insulin | Visit 1 (Baseline), Visit 3 (Week 12)
  Measured through plasma concentrations Unit/ml
Triglycerides | Visit 1 (Baseline), Visit 3 (Week 12)
  Plasma concentrations (mg/dl)
HDL (high-density lipoprotein)-cholesterol | Visit 1 (Baseline), Visit 3 (Week 12)
  Plasma concentrations (mg/dl)
LDL (low-density lipoprotein)-cholesterol | Visit 1 (Baseline), Visit 3 (Week 12)
  Plasma concentrations (mg/dl)
Total cholesterol | Visit 1 (Baseline), Visit 3 (Week 12)
  Plasma concentrations (mg/dl)
Waist circumference | Visit 1 (baseline), visit 2 (week 6), visit 3 (week 12)
  Unit: centimetres Measured with: ergonomic measuring tape
Hip circumference | Visit 1 (Baseline), Visit 2 (Week 6), Visit 3 (Week 12)
  Unit: centimetres Measured with: ergonomic measuring tape
Fat mass | Visit 1 (baseline), visit 2 (week 6), visit 3 (week 12)
  Unit: % Measured with: bioimpedance scan
Muscle mass | Visit 1 (Baseline), Visit 2 (Week 6), Visit 3 (Week 12)
  Unit: % Measured with: bioimpedance scan
Alanine aminotransferase | Visit 1 (Baseline), Visit 3 (Week 12)
  Measured through plasma concentrations: Unit: units/litre
Aspartate aminotransferase | Visit 1 (Baseline), Visit 3 (Week 12)
  Measured through plasma concentrations Units: units/litre
Bilirrubin | Visit 1 (Baseline), Visit 3 (Week 12)
  Measured through plasma concentrations Unit: mg/dl
Creatinin | Visit 1 (Baseline), Visit 3 (Week 12)
  Measured through plasma concentrations (mg/dl)
Urea | Visit 1 (Baseline), Visit 3 (Week 12)
  Measured through plasma concentrations (mg/dl)
Uric acid | Visit 1 (Baseline), Visit 3 (Week 12)
  Measured through plasma concentrations Unit: mg/dl
Hemoglobin | Visit 1 (Baseline), Visit 3 (Week 12)
  Plasma concentrations (g/dl)
Erithrocytes | Visit 1 (Baseline), Visit 3 (Week 12)
  Plasma concentrations (cel/mcl)
Leucocytes | Visit 1 (Baseline), Visit 3 (Week 12)
  Plasma concentrations (cel/mcl)
Thyroid-stimulating hormone (TSH) | Visit 1 (Baseline), Visit 3 (Week 12)
  Measured through plasma concentrations (mU/litre)
Dietary intake | Visit 1 (Baseline), Visit 3 (Week 12)
  24-h dietary recall and food frequency questionnaire
Physical activity level | Visit 1 (Baseline), Visit 3 (Week 12)
  Unit: MET-min per week Measured with: International Physical Activity Questionnaire (IPAQ)
  Low: Individuals who do not meet the criteria for Moderate or High categories.
  Moderate: Meeting one of the following criteria: (1) Three or more days of vigorous activity of at least 20 minutes per day. (2) Five or more days of moderate-intensity activity or walking of at least 30 minutes per day. (3) Five or more days of any combination of walking, moderate-intensity, or vigorous-intensity activities achieving a minimum of at least 600 MET-minutes per week.
  High: Meeting one of the following criteria: (1) Vigorous-intensity activity on at least 3 days accumulating at least 1500 MET-minutes per week. (2) Seven or more days of any combination of walking, moderate-intensity, or vigorous-intensity activities accumulating a minimum of at least 3000 MET-minutes per week.
Physical activity | Visit 1 (Baseline), Visit 3 (Week 12)
  Unit: Steps and time (hours) Measured with: ActivPAL accelerometers
Handgrip strength | Visit 1 (Baseline), Visit 3 (Week 12)
  Unit: Kilograms Measured with: Jamar plus dynamometer
Isometric Knee Extension Strength | Visit 1 (Baseline), Visit 3 (Week 12)
  Unit: Kilograms Measured with: Tindeq Progressor 200 dynamometer
Physical self-concept | Visit 1 (Baseline), Visit 3 (Week 12)
  Unit: points Measured with: Physical self-concept questionnaire (CAF)
  It consists of 36 items, grouped into 6 dimensions. The items are rated on a 5-point Likert-type scale, where 1 means false and 5 means true. The minimum and maximum scores per dimension are 6 and 30, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Fabian Lanuza, Temuco, Región de la Araucanía, Chile

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared due to confidentiality agreements with participants. Aggregate data will be included in scientific publications.

REFERENCES:
- [Derived] Lanuza F, Romero-Lopez C, Nova-Luna R, Cuyul-Vasquez I, Saez-Venegas M, Guzman N, Diaz-Velis L, Zamora-Ros R, Martinez-Huelamo M, Andres-Lacueva C. Effect of plant-based foods and (poly)phenol supplementation on gut-microbiota metabolism in participants with overweight or obesity and cardiometabolic risk: a study protocol for a single-blind, parallel and randomised controlled trial. BMJ Open. 2025 Sep 16;15(9):e105461. doi: 10.1136/bmjopen-2025-105461. PMID 40962336